CLINICAL TRIAL: NCT05936905
Title: A Controlled Clinical Trial of Group Acupuncture Therapy VS Chiropractor Group Therapy to Reduce Anxiety and Depression in People Living With HIV/AIDS (PLWH/A).
Brief Title: Acupuncture Therapy VS Chiropractor Group Therapy to Reduce Anxiety and Depression.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yo San University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Robert Hoffman, CEO/DEAN, Yo San University of Traditional Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YSU8232022
Record Dates: First submitted 2023-06-22; First posted 2023-07-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Anxiety Depression; HIV/AIDS
Keywords: Anxiety and depression; People living with HIV/AIDS (PLWH/A); Acupuncture; Chiropractor
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Anxiety Disorders; Depression | interventions — Acupuncture Therapy; Manipulation, Chiropractic

STUDY DESIGN:
Intervention Model Description: Staff members will administer the HADS, PHQ-9 and GAD-7 through a questionnaire. The scale is being administered to a convenience sample of 30 HIV/AIDs patients, divided into 15 samples of acupuncture treatment and 15 samples of chiropractor treatment, duration 3 months. Patients will complete questionnaire before and at the end of the treatments. Data to be collected includes socio-demographic. Symptoms of anxiety and depression are measured using the Hospital Anxiety and Depression Scale (HADS). The items are rated on 0, 1, 2, and 3 giving scores with minimum scores of 0 to 21. Scores on anxiety or depression subscales ranging from 0-7 are considered normal; 8-10 are considered cause for concern, borderline abnormal, and 11-21 are considered abnormal probable cases of anxiety or depression. The Patient Health Questionnaire 9-item(PHQ-9) if (score ≥9) significant mild depressive symptom and Generalized Anxiety Disorder 7-item (GAD-7) scale, if (score 8+) probable anxiety disorder.
Who Masked: Care Provider, Investigator
Masking Description: Single blind non randomized clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture therapy (Experimental): This study aims to compare acupuncture therapy administered one time per month
  Interventions: Other: Acupuncture
- Chiropractor therapy (Experimental): This study aims to compare chiropractic therapy administered one time per month
  Interventions: Other: Chiropractic

INTERVENTIONS:
Other: Acupuncture — Acupuncture 1 time per month
  Arms: Acupuncture therapy
Other: Chiropractic — Chiropractic 1 time per month
  Arms: Chiropractor therapy

SUMMARY:
This study aims to determine and compare acupuncture therapy and chiropractor group therapy to reduce anxiety and depression among HIV/AIDS patients at Being Alive, Los Angeles. In this controlled clinical trial, a total of 30 patients will be divided into two groups, 15 in the acupuncture therapy group, 15 in the chiropractor group therapy. The Hospital Anxiety and Depression Scale (HADS), The Patient Health Questionnaire 9-item (PHQ-9) and Generalized Anxiety Disorder 7- item scales (GAD-7) will be used as screening tools for depressive and anxiety symptoms respectively.

DETAILED DESCRIPTION:
In this study, the objectives are to determine and compare the prevalence of symptoms of depression and anxiety and find the most effective treatment method to assist patients in improving their quality of life utilizing holistic health treatments such as acupuncture and chiropractic to support their physical and mental health. Depression and anxiety are currently a major public health challenge worldwide especially during the Covid-19 pandemic. Approximately 280 million people within the world have depression, and over 700,000 people die due to suicide per annum (WHO, 2021). This depression and anxiety in PLWHAs can result in poor quality of life, and quality of work, school, and family life. Also, risky sexual behavior, the spreading of the virus, and at its worst, depression can result in suicide.

This controlled clinical trial will explore the treatment of acupuncture versus chiropractor care to seek out which treatment can help people living with HIV/AIDS (PLWH/A) to reduce depression and anxiety among PLWH/A patients in Being Alive, Los Angeles.

ELIGIBILITY:
Inclusion Criteria:

* single intervention only

Exclusion Criteria:

* chiropractic and acupuncture together

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 3 months
  Seven item questionnaire of each anxiety and depression. The items are rated on 0, 1, 2, and 3 giving scores with minimum scores of 0 to 21 maximum. Score interpretation on anxiety or depression subscales ranging from 0-7 considered non case, 8-10 considered possible case, and 11-21 considered probable case, which have been reclassified and relabeled as follows: 0-7 normal, 8-10 = mild, 11-15= moderate, and ≥16 = severe of anxiety or depression.
The Patient Health Questionnaire 9-item (PHQ-9) | 3 months
  Patient Health Questionnaire for depression, score interpretation. Severity. The developers report the following interpretive guidelines for the PHQ-9 as a severity measure: 1-4 no depression, 5-9 = mild de- pression, 10-14= moderate depression, 15-19 = moderately severe depression, and 20-27= severe depression.
Generalized Anxiety Disorder 7-item (GAD-7) | 3 months
  Anxiety Disorder 7-item, scoring Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate, and severe anxiety, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Yo San University, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No